# Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device Clinical Trial Protocol

Protocol Version and Date V1.1. 20250320

Clinical Research Unit Affiliated Hospital of Nantong University

Principal Investigator Prof. Lu Qi

Sponsor Affiliated Hospital of Nantong University

#### Confidentiality Statement

The information contained in the clinical protocol can only be provided to the investigator, other personnel involved in the clinical trial and the ethics committee. Except for the informed consent of the subjects, the information contained in this document shall not be disclosed to any third party not related to the clinical trial without the written consent of the sponsor.

# Table of contents

| List of abbreviations | 4 |
|---|---|
| Summary of the Trial Protocol | 5 |
| Text of the Trial Protocol | 9 |
| 1. Study information | 9 |
| 2. Background | 9 |
| 3. Study design | 10 |
| 3.1 Purpose | |
| 3.2 Selection of subjects 4. Study process | |
| 4.1 Test flow | 11 |
| 4.2 Subjects completion/withdrawal from the trial | |
| 6. Statistical analysis | 14 |
| 6.1 Sample size calculation | |
| 6.2 Methods of statistical analysis | |
| 7.1 Ethics Committee | 15 |
| 7.2 Informed consent form 8. Definition of adverse events and response measures | |
| 8.1 Adverse events | 15 |
| 8.2 Serious Adverse Events | |
| 8.4 Expected adverse reactions | 17 |
| 8.5 Duration of follow-up after adverse events 8.6 Security incident audits | |
| Annex I: CHA2DS2-VASc Score for Nonvalvular Atrial Fibrillation Stroke Risk | |
| Annex II: HAS-BLED Score | 22 |
| Annex III: PASS Principles | 23 |
| Annex IV: Atrial Fibrillation Effect on Quality-of-Life questionnaire (Al | _ / |
| | 25 |

## List of abbreviations

| No. | abbreviations | the complete English alphabet |
|-----|---------------|------------------------------------------|
| 1 | NMPA | National Medical Products Administration |
| 2 | EC | Ethics Committee |
| 3 | ICF | Informed Consent Form |
| 4 | CRF | Case Report Form |
| 5 | SOP | Standard Operating Procedure |
| 6 | LAA | Left Atrial Appendage |
| 7 | ТТЕ | Transthoracic Echocardiography |
| 8 | TEE | Transesophageal Echocardiography |
| 9 | LVEF | Left Ventricular Ejection Fraction |
| 10 | LAFF | Left Atrial Flow Fraction |
| 11 | DSA | Digital Subtraction Angiography |
| 12 | AF | Atrial Fibrillation |
| 13 | AE | Adverse Event |
| 14 | MAE | Major Adverse Event |
| 15 | SAE | Serious Adverse Event |
| 16 | DRT | Device Related Thrombosis |
| 17 | ICE | Intracardiac Echocardiography |
| 18 | EDC | Electronic Data Capture System |
| 19 | BMI | Body Mass Index |
| 20 | LAAO | Left Atrial Appendage Occlusion |

# **Summary of the Trial Protocol**

| Test Name | Evaluation of the Safety and Efficacy of Catheter Ablation After Left Atric |
|---|---|
| l'est Name | Appendage Occlusion with the WATCHMAN FLX Device |
| Sponsor | Department of Cardiology, Affiliated Hospital of Nantong University |
| Principal | Professor Lu Qi |
| Investigator | Professor Lu Qi |
| | 1. Main Purpose: |
| | To evaluate the safety and efficacy of catheter ablation performed one month |
| | after WATCHMAN FLX left atrial appendage occlusion (LAAO) in patients |
| | with non-valvular atrial fibrillation(AF). |
| Purpose of the test | 2. Secondary Purpose: |
| | To investigate the impact of a two-surgery sequential treatment regimen on the |
| | recurrence rate of atrial fibrillation, the incidence of stroke, and the quality of |
| | life of patients, and to provide evidence-based support for decision-making in |
| | the clinical application of combined therapy. |
| | Patients diagnosed with non-valvular AF who are scheduled to undergo |
| Trial Population | sequential LAAO using the WATCHMAN FLX device and catheter-based |
| | ablation. |
| | This study is a prospective, single-arm, multicenter clinical trial designed to |
| | evaluate the safety and efficacy of catheter ablation performed one month after |
| | LAAO with the WATCHMAN FLX device. Approximately 210 patients with |
| | non-valvular AF who meet the indications for both transcatheter LAAO and |
| | catheter ablation will be enrolled across 10 research centers in China. The |
| | study procedures are outlined as follows:: |
| | 1. Patient Screening and Enrollment: Eligible patients will undergo |
| Trial Design | elective LAAO with the WATCHMAN FLX device (first procedure) |
| | after signing the informed consent form (ICF). |
| | 2. Postoperative Management: Following the LAAO with the |
| | WATCHMAN FLX device, patients will undergo standard |
| | anticoagulation therapy for one month. If transesophageal |
| | echocardiography (TEE) reveals no device-related thrombosis (DRT) |
| | or residual flow >5 mm, the patient will undergo catheter ablation for |
| | atrial fibrillation (second procedure) one month after the initial LAAO. |

| Evaluation of the Safety and Eff | icacy of Ca | atheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device |
|---|---|---|
| | 3. | Follow-up: Baseline patient data will be collected prior to the first |

procedure. Follow-up visits will occur within 7 days post-LAAO or at discharge, and at 1 month (i.e., time of the second procedure), 3 months, and 12 months post-procedure. Follow-up will focus on device endothelialization at 12 months, recurrence of atrial fibrillation, and

occurrence of related complications.

Postoperative Medication Management Strategy:

Patients will receive anticoagulation therapy for 1 month following LAAO with the WATCHMAN FLX device. If no thrombosis or significant residual flow is detected, catheter ablation for atrial fibrillation will be performed. After the ablation procedure, anticoagulation therapy will be continued for an additional 2 months. Antiarrhythmic drugs (AADs) may be used within 90 days post-ablation in accordance with AF management guidelines.

The success rate of complete left atrial appendage (LAA) closure within 12 **Primary endpoint** months following LAAO with the WATCHMAN FLX device, as assessed by LAA computed tomography angiography (CTA).

#### **Safety Endpoints:**

Incidence of procedure-related complications and adverse events within 30 days after LAAO and radiofrequency ablation, including rates of pericardial effusion, access site complications, vascular complications, and infections. The incidence of procedure-related complications and adverse events within 12 months following LAAO and radiofrequency ablation will be evaluated. These include major bleeding events (defined as those requiring blood transfusion or surgical intervention), cardiac tamponade, systemic embolism (including ischemic stroke and other embolic events), device-related thrombosis (DRT), new or enlarged peri-device leak (PDL, defined as >5 mm), acute postoperative left heart failure, and rehospitalization.

### Secondary endpoint

#### **Efficacy Endpoints:**

- 1. Treatment success rate within 3 months after radiofrequency ablation (Early recurrence): No recurrence of atrial arrhythmias ≥30 seconds.
- 2. Treatment success rate between 4 to 12 months after ablation (Late recurrence): No recurrence of atrial arrhythmias ≥30 seconds during this period.
- 3. Incidence of stroke within 12 months following LAAO: No occurrence of stroke.

| Evaluation of the Safety and Eff | icacy of Cath | eter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device |
|---|---|---|
| Evaluation of the Statety and Eff | | Quality of life improvement at 12 months measured by the Atrial |
| | F | Fibrillation Effect on Quality-of-Life (AFEQT) questionnaire: |
| | I | mprovement in quality-of-life score from baseline to 12 months |
| | f | following index ablation or AAD treatment, with a possible score |
| | r | ange of 20 to 140 (higher scores indicate worse outcomes). |
| | 1) | Age ≥18 years with a diagnosis of nonvalvular AF; |
| | 2) | Eligible for indications for treatment with WATCHMAN FLX |
| Endam Cuidania | | LAAO and transcatheter atrial fibrillation ablation; |
| Entry Criteria | 3) | Preoperative imaging evaluation showed that the LAA anatomy was |
| | | suitable for WATCHMAN FLX device implantation; |
| | 4) | Patients agreed to participate in the study and signed an ICF. |
| | Patients | meeting any of the following criteria were not eligible for this study: |
| | 1) | Presence of valvular heart disease or other structural heart disease |
| | that caus | ses atrial fibrillation; |
| | 2) | Preoperative detection of LAA thrombus or acute thrombotic event; |
| | 3) | The patient has a severe bleeding tendency or a recent major |
| <b>Exclusion criteria</b> | bleeding | g event (e.g. gastrointestinal hemorrhage, cerebral hemorrhage, etc.); |
| | 4) | Patients who are unable to complete postoperative follow-up (e.g. |
| | life expe | ectancy less than 1 year or poor compliance); |
| | 5) | Other serious diseases (e.g. liver and kidney failure, active |
| | infection | ns, etc.) detected on preoperative examination; |
| | 6) | Women who are pregnant or breastfeeding. |
| | 1. 8 | Sample size calculation: |
| | The sam | ple size was calculated based on the primary endpoint. The primary |
| | endpoint | t of this study was "12-month rate of complete closure of the block |
| | after W | ATCHMAN FLX LAAO (CT assessment)." |
| | Hypothe | sized target incidence P0= 74.3% and test incidence P1= 84.3%. The |
| statistical analysis | significa | ance level $\alpha = 0.05$ (one-sided) and test efficacy 1- $\beta = 80\%$ were |
| | calculated to be 200 cases able to fulfill the hypothesis test. Considering the | |
| | 5% shed | ding rate, the total sample size was 210 cases. |
| | 2. I | Descriptive Statistics: |
| | Patient b | paseline characteristics (e.g. age, sex, history of AF) were expressed |
| | as mean: | ± standard deviation or median (quartiles) for continuous variables, |

and frequency and percentage for categorical variables.

#### 3. Primary endpoint analysis:

The 12-month complete closure rate of the WATCHMAN FLX device was characterized by point estimates and their 95% confidence intervals and tested against the target value of  $P_0 = 74.3\%$  in a one-sample hypothesis test ( $\alpha = 0.05$ ).

#### 4. Secondary endpoint analysis:

Safety events (e.g.pericardial effusion, puncture site complications) were described by incidence rates and their 95% confidence intervals were calculated. Changes in quality of life were analyzed by chi-square test or paired t-test for time effects.

#### **Text of the Trial Protocol**

#### 1. Study information

Name of Sponsor: Affiliated Hospital of Nantong University

Principal Investigator: Prof. Lu Qi

#### 2. Background

Atrial fibrillation (AF) is one of the most common persistent arrhythmias in clinical practice, and its prevalence increases significantly with age, posing a serious threat to public health globally [1]. One of the most serious complications in patients with AF is thromboembolic events, especially cardioembolic stroke. Cardioembolic strokes due to AF account for 20-30% of all strokes and are associated with significantly higher rates of mortality and disability in post-stroke patients [2]. Studies have shown that approximately 90% of blood clots in patients with nonvalvular atrial fibrillation originate from the left atrial appendage (LAA) [3]; therefore, preventing stroke by isolating the LAA from the atria has become an important strategy in the management of patients with AF, a surgical procedure known as left atrial appendage occlusion (LAAO) [4]. Furthermore, international and national guidelines for arrhythmia management state that rhythm control and stroke prevention are equally important in patients with AF. Although LAAO has been shown to be effective in reducing the risk of stroke associated with AF [5], it does not address the arrhythmia of the patient. In contrast, catheter ablation is one of the most effective treatments for rhythm control, and has been shown in several randomized controlled trials (RCTs) to significantly improve sinus rhythm maintenance and quality of life in patients with AF [6-9]. These studies have shown that catheter ablation is the method of choice for rhythm control in patients with paroxysmal AF, with better long-term outcomes compared with pharmacologic therapy. To address rhythm control and stroke prevention in patients with AF in an integrated manner, combining catheter ablation and LAAO is a feasible and promising therapeutic strategy. Catheter ablation aims to restore sinus rhythm by intervening in the triggering mechanism of AF, whereas LAAO reduces the risk of stroke by isolating the main site of thrombus formation. The combination of the two surgical approaches not only improves the maintenance of sinus rhythm in patients, but also significantly reduces the risk of stroke and all-cause mortality [10].

Currently, the use of combinations of these two procedures is increasing in clinical practice. Some studies and expert consensus suggest that the goal of integrated therapy can be achieved by "one-stop surgery" (performing both catheter ablation and LAAO in a single operation) or staged surgery (performing one procedure before the other) [11].

Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device However, there are no uniform conclusions regarding the optimal sequence of procedures. Some studies have shown that concurrent "one-stop" surgery may reduce hospitalization time, surgical risk, and patient financial burden [12], while staged surgery allows physicians to better assess outcomes after the initial surgery and reduces the overall surgical risk to the patient [13].

The 2021 expert consensus on the management of atrial fibrillation in China made a class IIb recommendation for "one-stop surgery", suggesting that for some patients with nonvalvular AF who have indications for both catheter ablation and LAAO, it is reasonable to perform LAAO at the same time as catheter ablation. Nevertheless, there is a lack of trials to validate the advantages and disadvantages of different procedural sequences in terms of safety and efficacy.

Therefore, the aim of this study was to evaluate the safety and efficacy of transcatheter AF ablation 1 month after WATCHMAN FLX LAAO, to provide an evidence-based medical rationale for optimizing the comprehensive management of patients with AF, and to further explore the optimal combined strategy of the two surgical approaches in patients with nonvalvular AF.

#### 3. Study design

#### 3.1 Purpose

#### 3.1.1 Main Purpose

To evaluate the safety and efficacy of catheter ablation performed one month after WATCHMAN FLX left atrial appendage occlusion (LAAO) in patients with non-valvular atrial fibrillation (AF).

#### 3.1.2 Secondary Purpose

To investigate the impact of a two-surgery sequential treatment regimen on the recurrence rate of atrial fibrillation, the incidence of stroke, and the quality of life of patients, and to provide evidence-based support for decision-making in the clinical application of combined therapy.

#### 3.2 Selection of subjects

#### 3.2.1 Entry Criteria

- 1) Age  $\geq$ 18 years with a diagnosis of nonvalvular AF;
- 2) Eligible for indications for treatment with WATCHMAN FLX LAAO and transcatheter atrial fibrillation ablation;
- 3) Preoperative imaging evaluation showed that the LAA anatomy was suitable for WATCHMAN FLX device implantation;
- 4) Patients agreed to participate in the study and signed an ICF.

#### 3.2.2 Exclusion criteria

Patients meeting any of the following criteria were not eligible for this study:

- 1) Presence of valvular heart disease or other structural heart disease that causes atrial fibrillation;
  - 2) Preoperative detection of LAA thrombus or acute thrombotic event;
- 3) The patient has a severe bleeding tendency or a recent major bleeding event (e.g. gastrointestinal hemorrhage, cerebral hemorrhage, etc.);
- 4) Patients who are unable to complete postoperative follow-up (e.g. life expectancy less than 1 year or poor compliance);
- 5) Other serious diseases (e.g. liver and kidney failure, active infections, etc.) detected on preoperative examination;
  - 6) Women who are pregnant or breastfeeding.

#### 4. Study process

#### 4.1 Test flow

| Visiting | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| time Visiting Program | screening<br>period | intraoperative<br>(LAAO) | LAAO postoperative to discharge or 7 days postoperative | 1 month after<br>surgery<br>(ablation) | Post-ablation to<br>discharge or 7<br>days<br>post-procedure | 3 months after<br>surgery | 1 year after<br>surgery |
| informed consent | $\blacktriangle^1$ | | | | | | |
| Inclusion/exclusi<br>on criteria | <b>A</b> | | | | | | |
| Demographic information | <b>A</b> | | | | | | |
| Medical history <sup>2</sup> | <b>A</b> | | | | | | |
| Surgical information <sup>3</sup> | | <b>A</b> | | <b>A</b> | | | |
| CHA <sub>2</sub> DS <sub>2</sub> -VASc<br>score | <b>A</b> | | | | | | |
| HAS-BLED score | <b>A</b> | | | | | | |
| MRS Rating Scale 4 | Δ | | Δ | | Δ | Δ | Δ |
| routine blood test | <b>A</b> | | <b>A</b> | | <b>A</b> | <b>A</b> | <b>A</b> |
| Renal function <sup>5</sup> | <b>A</b> | | <b>A</b> | | <b>A</b> | <b>A</b> | <b>A</b> |
| Coagulation INR | <b>A</b> | | • | | <b>A</b> | Δ | Δ |

Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device

| TEE | Δ | | Δ | | Δ | Δ | Δ |
|---|---|---|---|---|---|---|---|
| CT | Δ | | Δ | | Δ | Δ | <b>A</b> |
| 12-lead electrocardiogram <sup>6</sup> | <b>A</b> | | <b>A</b> | | <b>A</b> | <b>A</b> | <b>A</b> |
| Combined medication 8 | <b>A</b> | | <b>A</b> | | <b>A</b> | <b>A</b> | <b>A</b> |
| adverse event | <b>A</b> | <b>A</b> | <b>A</b> | <b>A</b> | <b>A</b> | <b>A</b> | <b>A</b> |

Remarks:

- 1. For the active collection of information, the examination items were completed according to the needs of patients' diagnosis and treatment evaluation and clinical research;  $\triangle$  For the selective collection of information, the researcher judged and chose to complete these examination items according to the actual health status of the patients, and this study did not intervene/require the patients to complete these examination items.
- 2. Medical history: including past medical history, family history, history of atrial fibrillation, personal history, medication history, surgical history, history of hypertension, diabetes mellitus, coronary artery disease, heart failure, peripheral vascular disease, history of hepatic and renal disease, stroke or systemic embolism, and cardiovascular-related surgery
- 3. Surgical information: intraoperative imaging such as DSA, other intraoperative information such as anesthesia, anticoagulant dosage, perioperative surgical complications, surgical approach, etc.
- 4. Evaluate when a neurological event occurs
- 5. Renal function: creatinine, creatinine clearance
- 6. 12-lead electrocardiogram: the most recent occurrence was recorded during both the screening and follow-up periods.
  Combined medications: record of anticoagulants, antiplatelet agents, antihypertensive agents, lipid-lowering agents, hypoglycemic agents, and medications to treat surgical complications.

#### 4.2 Subjects completion/withdrawal from the trial

#### 4.2.1 Completion of studies

Patients met inclusion/exclusion criteria and signed ICF until completion of 1 year of follow-up.

#### 4.2.2 Termination of treatment

Patients have the right to withdraw from the study at any time without any reason and their subsequent treatment will not be affected in any way by this. Subjects should discontinue study treatment if any of the following occurs:

- (1) Significant protocol violations (including poor adherence, failure to meet inclusion criteria or meeting exclusion criteria for enrollment, etc.) as confirmed by the principal investigator (PI);
  - (2) Serious procedure-related complications during percutaneous LAAO;
- (3) Patients who are no longer suitable for continued participation in the study due to adverse events for patient safety reasons;
  - (4) The patient refuses to participate or refuses to continue to participate in this study;
  - (5) Pregnancy.

#### 4.2.3 Exit trial

This subject will be withdrawn from the trial for the following reasons:

- (1) Death;
- (2) Lost visits;
- (3) Withdrawal of ICF.

Subjects who terminate or withdraw early from the study are required to be contacted by research center staff making every effort to determine the reason for early termination or withdrawal and the presence of any adverse events. Subjects who terminate or withdraw early from the study need to be thoroughly evaluated at the final visit and documented as thoroughly as possible. The reason for early termination or withdrawal from the study, the date, and the final evaluation must be documented in the study materials.

# 5. Data management and statistical analysis plan, information confidentiality plan

A clinical trial summary report will be written based on the statistical analysis report. The investigator maintains all study materials, including confirmation of all participating subjects (able to effectively verify different recorded information, such as original hospital records), all original informed consent forms signed by the patient, and all case observation forms. The investigator will keep the information about the subjects closely until its final destruction, during which time it will not continue to use or disclose the information.

Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device However, in the rare cases listed below, the investigator will continue to use or disclose information about a subject even if the subject has withdrawn from the study or the study has been completed. These situations include: when the removal of the subject's information would affect the scientific validity of the results of the study or the evaluation of the safety of the data; to provide some limited information for research, teaching, or other activities (this information will not include names, identification numbers, or other personally identifiable information); when government regulators need to oversee the study, they will ask to see all of the information about the study, which will also include information about the subject's information about their participation in the study at that time.

#### 6. Statistical analysis

#### 6.1 Sample size calculation

The sample size was calculated based on the primary endpoint. The primary endpoint of this study was "12-month rate of complete closure of the block after WATCHMAN FLX LAAO (CT assessment)".

Assuming that P0is the target incidence rate and P1is the trial incidence rate, P0was set to 74.3% (95% confidence interval: 65.9% ~ 82.7%) based on the literature reports\*and expert recommendations, the hypothesis testing was as follows:

$$H0: P1 \leq 0.743$$

H1: 
$$P1 > 0.743$$

A P1of 84.3% was set, significance level  $\alpha = 0.05$  (one-sided), and test efficacy 1- $\beta = 80\%$ . According to the sample size formula, 200 patients were needed in a single group to fulfill the statistical requirements. Considering a 5% loss-to-follow-up rate, the total sample size was set at 210 cases.

\*Yoon SH, Amoah JK, Galo J, Dallan LAP, Arruda M, Rashid I, Rajagopalan S, Filby SJ. Incidence, progression, and predictors of left atrial appendage sealing after Watchman FLX device implantation with computed tomographic assessment. Catheter Cardiovasc Interv. 2024
May; 103(6):995-1003. doi: 10.1002/ccd.31044. Epub 2024 Apr 25. PMID: 38662126.

#### **6.2** Methods of statistical analysis

#### 6.2.1 Analysis sets

The Intent-to-Treat (ITT) set includes all participants who signed the ICF and meet inclusion/exclusion criteria.

#### 6.2.2 Data analysis

Patient baseline characteristics (e.g. age, sex, history of atrial fibrillation) were expressed as mean± standard deviation or median (quartiles) for continuous variables, and frequency and percentage for categorical variables.

Primary endpoint analysis:

Analyses of the primary endpoints will be performed based on mITT, with the 12-month complete closure rate of the WATCHMAN FLX device described by point estimates and their 95% confidence intervals, and a one-proportional hypothesis test ( $\alpha = 0.05$ ) against a target value of  $P_0 = 74.3\%$ .

Secondary endpoint analysis:

Safety events (e.g. pericardial effusion, puncture site complications) were described by incidence rates and their 95% confidence intervals were calculated. Changes in quality of life were analyzed by chi-square test or paired t-test for time effects.

#### 7. Ethical requirements and informed consent form

#### 7.1 Ethics Committee

Prior to the clinical study, the investigator is required to submit the clinical study protocol, informed consent and other relevant documents to the ethics committee of the hospital where the unit responsible for the clinical study is located. The clinical study can only be started after obtaining the approval of the ethics committee (sub-centers can also start the clinical study after accepting the ethics of the group leader center). Any modification of the study protocol must be approved by the Ethics Committee before implementation. Serious adverse events in the course of the clinical study should be submitted to the Ethics Committee in writing in a timely manner (each center will report according to the ethical requirements of each center, and back up to the group leader unit at the same time).

#### 7.2 Informed consent form

Prior to enrollment in this study, the investigator must inform the subjects and their relatives about the details of the clinical study, including the content of the study, the purpose of the study, the expected efficacy, possible adverse events and countermeasures. Subjects will be enrolled only after they fully understand the study and sign an informed consent form. The informed consent form will be signed in duplicate by the study physician and the subject himself/herself or his/her legal representative, and each party will keep a copy.

#### 8. Definition of adverse events and response measures

#### 8.1 Adverse events

#### 8.1.1 Definition of adverse events

An adverse event is an adverse medical condition or a worsening of a pre-existing medical condition that occurs after the implantation of an investigational device or during the course of treatment, whether or not there is a causal relationship between the condition and the investigational device. This adverse medical condition can be a symptom (e.g., nausea, chest pain), sign (e.g., tachycardia, hepatomegaly), or an abnormal test result (e.g., laboratory result, electrocardiogram). In a clinical study, an AE can encompass an adverse medical condition that occurs at any time, including the introductory or washout period, even when no study treatment is given.

#### 8.1.2 Determination of severity of adverse events

Mild: Does not interfere with daily activities;

Moderate: interferes with daily activities;

Severe: Loss of ability to perform daily activities.

#### 8.1.3 Response to adverse events

All adverse events occurring during the study period must be faithfully recorded in the Adverse Event Form, and the investigator should give targeted treatment for the adverse event and follow up until the symptoms have disappeared or stabilized.

#### **8.2 Serious Adverse Events**

#### 8.2.1 Definition of serious adverse events

A serious adverse event is defined as an AE that occurs within any study phase (i.e. introductory, treatment, washout, follow-up) that meets 1 or more of the following criteria.

- Lead to death
- Immediately life-threatening
- Subject hospitalization or extension of existing hospitalization is required
- Cause permanent or significant disability or dysfunction
- Cause congenital malformations or birth defects
- Significant medical events that may jeopardize the health of the subject or require medical intervention to avoid the above outcomes

#### 8.2.2 Reporting process

In the event of a serious adverse event in a clinical trial, the investigator shall immediately take appropriate therapeutic measures for the subject, and at the same time report in writing to the drug clinical trial management department of the clinical trial organization to which it belongs, and by which the sponsor shall be notified in writing. The clinical trial management department shall, within 24 hours, report in writing to the appropriate ethics committee as well as the food and drug supervision and management

Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device department of the province, autonomous region and municipality directly under the central government where the clinical trial organization is located and the competent department of health and family planning. In the case of a death, the clinical trial organization and the investigator shall provide the ethics committee and the sponsor with all the information required.

#### **8.3 Unintended Adverse Reactions**

Unintended adverse reactions are defined as serious adverse reactions affecting health, safety, or any life-threatening, death-causing problems or deaths arising from or associated with the investigational device, which were not identified in the prior study plan or application with respect to their severity or occurrence; or any other unintended serious device-related problems associated with patient rights, safety.

During the study, the investigator must, as far as possible, refer any occurrence of unintended adverse reactions to the Principal Investigator and the Ethics Committee. Serious adverse reactions were reported within 24 hours. The Principal Investigator and Ethics Committee inform the investigator of any unintended device adverse reactions that occur.

#### 8.4 Expected adverse reactions

The following anticipated complications may result from the occluder or antithrombotic medications:

1, Device related thrombosis 2, Ischemic stroke 3, Pericardial effusion 4, Hemorrhagic stroke 5, Cardiac tamponade 6, Nuisance bleeding 7, Hemorrhage 8, Death

#### 8.5 Duration of follow-up after adverse events

All adverse events are to be followed until resolved or until a stable clinical endpoint is achieved

#### 8.6 Security incident audits

To ensure the safety of subjects during the conduct of the study, the safety of the clinical trial will be assessed by analyzing and reviewing major safety events at regular intervals during the conduct of the study. Given that all-cause mortality, ischemic stroke, and major bleeding events are the most relevant adverse events related to device or procedure safety, the focus will be on monitoring and evaluating these three types of events. Once the number of subjects with safety events reaches or exceeds the expected number of cases, safety investigations and appropriate treatment measures will be triggered.

#### **References:**

- Hindricks G, Potpara T, Dagres N, et al. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). *Eur Heart J*. 2021;42(5):373-498. doi:10.1093/eurheartj/ehaa612
- Meschia JF, Bushnell C, Boden-Albala B, et al. Guidelines for the primary prevention of stroke: a statement for healthcare professionals from the American Heart Association/American Stroke Association. *Stroke*. 2014;45(12):3754-3832. doi:10.1161/STR.00000000000000046
- 3. Blackshear JL, Odell JA. Appendage obliteration to reduce stroke in cardiac surgical patients with atrial fibrillation. *Ann Thorac Surg.* 1996;61(2):755-759. doi:10.1016/0003-4975(95)00887-X
- Holmes DR, Kar S, Price MJ, et al. Prospective randomized evaluation of the WATCHMAN Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. *J Am Coll Cardiol*. 2014;64(1):1-12. doi:10.1016/j.jacc.2014.04.029
- Reddy VY, Sievert H, Halperin J, et al. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. *JAMA*. 2014;312(19):1988-1998. doi:10.1001/jama.2014.15192
- Wazni OM, Dandamudi G, Sood N, et al. Cryoballoon ablation as initial therapy for atrial fibrillation. N Engl J Med. 2021;384:316–24. doi:10.1056/NEJMoa2029554
- Cosedis Nielsen J, Johannessen A, Raatikainen P, et al. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation. N Engl J Med. 2012;367:1587–95. doi:10.1056/NEJMoa1113566
- Morillo CA, Verma A, Connolly SJ, et al. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of paroxysmal atrial fibrillation (RAAFT-2): a randomized trial. *JAMA*. 2014;311:692–700. doi:10.1001/jama.2014.467
- 9. Kuniss M, Pavlovic N, Velagic V, et al. Cryoballoon ablation vs. antiarrhythmic drugs: first-line therapy for patients with paroxysmal atrial fibrillation. *Europace*. 2021;23:1033-41. doi:10.1093/europace/euab029
- 10. Osmancik P, Herman D, Neuzil P, et al. Left atrial appendage closure versus direct oral anticoagulants in high-risk patients with atrial fibrillation. *J Am Coll Cardiol*. 2020;75(25):3122-3135. doi:10.1016/j.jacc.2020.04.067

- 11. Gianni C, Mohanty S, Trivedi C, et al. Two-staged hybrid surgical ablation and catheter ablation for the treatment of persistent and long-standing persistent atrial fibrillation. *J Am Coll Cardiol EP*. 2016;2(4):379-386. doi:10.1016/j.jacep.2016.01.024
- 12. Basu-Ray I, Liu J, Raghunathan D, et al. Safety and feasibility of one-stop hybrid epicardial-endocardial ablation and left atrial appendage closure for atrial fibrillation. *Heart Rhythm*. 2021;18(1):89-97. doi:10.1016/j.hrthm.2020.08.008
- Ellis CR, Sobieszczyk P. Left atrial appendage occlusion and atrial fibrillation ablation: a comprehensive approach. *Curr Cardiol Rep.* 2020;22(11):138. doi:10.1007/s11886-020-01370-2

#### Researcher's statement

I agree::

- 1. The clinical trial was conducted in strict accordance with the requirements of the Declaration of Helsinki, current Chinese regulations and the trial protocol.
- 2. The investigator writes a summary report of the clinical trial based on the statistical analysis report.
- 3. Test medical devices are used only for this clinical trial, and complete and accurate records of the receipt and use of test medical devices are kept in the course of the clinical trial.
- 4. Strictly fulfill the terms of the clinical trial contract/agreement signed by all parties. I have read the clinical trial protocol in its entirety, including the above statement, and I agree with all of the above.

| R | Researcher's opinion |
|---|----------------------|
| | ignature:<br>Date |

| Evaluation of the Safety and Efficacy of Catheter Ablation Following Left Atrial Appendage Occlusion Using the WATCHMAN FLX Device | |
|---|---|
| | Opinions of Medical Device Clinical Trial Organizations |
| | Signature (stamp) |
| | Data |
| | Date |

# Annex I: CHA<sub>2</sub>DS<sub>2</sub>-VASc Score for Nonvalvular Atrial Fibrillation Stroke Risk

| risk factor | Scoring (points) |
|-----------------------------------------------------------|------------------|
| Congestive heart failure/left ventricular dysfunction (C) | 1 |
| Hypertension (H) | 1 |
| Hypertension (H) | 2 |
| Diabetes (D) | 1 |
| Stroke/TIA/thromboembolism history (S) | 2 |
| Vascular disease history (V) | 1 |
| Age 65-74 (A) | 1 |
| Sex (Female, Sc) | 1 |
| maximum | 9 |

## **Annex II: HAS-BLED Score**

| Clinical features | Scoring<br>(points) |
|------------------------------------------------------|---------------------|
| Hypertension (H) | 1 |
| Abnormal liver and kidney function (1 point each, A) | 1 or 2 |
| Stroke(S) | 1 |
| Bleeding (B) | 1 |
| INR values are volatile (L) | 1 |
| Elderly (e.g. age >65 years, E) | 1 |
| Drugs or alcoholism (1 point each, D) | 1 |
| maximum | 9 |

# **Annex III: PASS Principles**

| | The shoulder of the earlyder is located at the strial annuadors ananing |
|---|---|
| | The shoulder of the occluder is located at the atrial appendage opening. |
| | "Three-position" angiography can be performed under X-ray fluoroscopy to |
| | check the positional relationship between the upper and lower edges of the |
| | occluder and the left atrial appendage opening. It is recommended that the |
| Position | height of the shoulder exposure be controlled within 1/3 of the occluder |
| | diameter. The shoulder exposure is usually adjusted at CAU20°+RAO0°-45° |
| | to clearly display the tangent position of the atrial side umbrella surface of |
| | the occluder, and the result is consistent with the corresponding angle of |
| | TEE. |
| | Slightly unscrew the hemostatic valve, withdraw the outer sheath about 2 cm |
| | away from the occluder umbrella, pull the release handle back 1.0-1.5 cm |
| | with moderate force, and release it immediately. There is obvious pulling |
| | resistance in this process. Under X-ray fluoroscopy, it is observed that the |
| | occluder and the atrial appendage wall move synchronously, and the |
| Anchor | occluder rebounds significantly after pulling, and there is no position change |
| | (contrast agent can be injected at the same time), and the device is stable. |
| | When the stability of the occluder is in doubt, it can be pulled again for |
| | verification. It is easier to judge the position change of the occluder by |
| | pulling at the tangent position of the side umbrella. |
| | The compression ratio is measured under X-ray fluoroscopy. Exposure can |
| | be performed in the right foot or right shoulder position (adjusted to the |
| | tangent position of the occluder), and the maximum diameter of the occluder |
| | is measured to calculate the compression ratio. The compression ratio is |
| Size | calculated as follows: (original size - expanded diameter) / original size × |
| | 100%, and the recommended value is 10% to 30%. At LAO 40°-50°, the |
| | entire umbrella surface on the atrial side of the occluder can be observed, and |
| | the maximum diameter can be measured through the center connection cap to |
| | calculate the compression ratio. |
| | Determine whether PDL exists after implantation of the occluder. |
| | "Three-position" angiography can be performed under X-ray fluoroscopy. |
| Seal | During angiography, check the positional relationship between the edge of |
| | the occluder and the atrial appendage orifice, and pay attention to whether |

contrast agent enters the left atrial appendage from around the occluder. If PDL is ≥3mm, adjust the position of the occluder or replace the occluder.

# Annex IV: Atrial Fibrillation Effect on Quality-of-Life

# questionnaire (AFEQT)

| Atrial Fibrillation Effect on | □No □Yes |
|---|---|
| Quality-of-Life questionnaire (AFEQT) | IF yes,please complete the AFEQT |
| In order to better understand the impact of AF on your health-related quality of life, we would like to | |
| ask you to answer the following questions and tick the appropriate box! | |
| (1) Palpitations: Panic, rapid heartbeat ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ 5 ☐ 6 ☐ Extremely | |
| (2) Irregular heartbeat | |
| $\square$ Not at all $\square 1 \square 2 \square 3 \square 4 \square 5 \square 6 \square$ Extremely | |
| (3) Dizziness and blurred vision ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ 5 ☐ 6 ☐ Extremely | |
| (4) Chest tightness, chest pain ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ 5 ☐ 6 ☐ Extremely | |
| (5) Worried that atrial fibrillation may strike at any time | |
| $\square$ Not at all $\square$ 1 $\square$ 2 $\square$ 3 $\square$ 4 $\square$ 5 $\square$ 6 $\square$ Extremely | |
| <ul> <li>(6) Worry that atrial fibrillation will worsen the disease in the long run.</li> <li>□ Not at all □1 □2 □3 □4 □5 □6 □ Extremely</li> </ul> | |
| (7) Concerns about side effects of dru ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ | lgs<br>]5 □6 □ Extremely |
| (8) Concerns about interventional procedures such as radiofrequency ablation, surgery, implantation of | |
| pacemaker Not at all 1 2 3 4 | ]5 □6 □ Extremely |
| (9) Worried about the side effects of | anticoagulant drugs, such as nosebleeds, bleeding gums when |
| brushing teeth, heavy bleeding or bru Not at all 1 2 3 4 | |
| (10) Fear that treatment will affect da Not at all 1 2 3 4 | ily life 5 \( \sum 6 \subseteq \) Extremely |
| (11) Recreation, leisure, sports, abilit ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ | |
| (12) Ability to get along with family members and do things together ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ 5 ☐ 6 ☐ Extremely | |
| (13) Limitations on mobility due to p Not at all 1 2 3 4 5 | erceived fatigue |
| (14) Limitations on mobility due to sl | - — — · |
| $\square$ Not at all $\square 1 \square 2 \square 3 \square 4 \square$ | |
| | ]5 □6 □ Extremely |
| (16) Go fast ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ | 5 □ 6 □ Extremely |
| | limbing stairs at a brisk pace without stopping for a break 5 \( \subseteq 6 \) Extremely |
| (18) Strenuous activities such as lifting heavy furniture, running, and strenuous sports such as | |
| squash/tennis/swimming/basketball. Not at all 1 2 3 4 5 6 Extremely | |
| (19) Effectiveness of current therapeutic measures to control housing fibrillation ☐ Not at all ☐ 1 ☐ 2 ☐ 3 ☐ 4 ☐ 5 ☐ 6 ☐ Extremely | |
| (20) Effectiveness of therapeutic measures in relieving symptoms associated with atrial fibrillation Not at all 1 2 3 4 5 6 Extremely | |